CLINICAL TRIAL: NCT03107442
Title: Effects of an Aerobic Exercise Intervention Program on Arterial Stiffness and Inflammation in Women With Systemic Lupus Erythematosus
Brief Title: Exercise and Arterial Stiffness in Systemic Lupus Erythematosus
Acronym: EJERCITALES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, José Antonio Vargas Hitos, José A. Vargas-Hitos, MD, PhD, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-0525-2016
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Arterial stiffness; Markers of Inflammation; Exercise; Physical fitness; Cardiovascular risk; Autoimmune diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity; Autoimmune Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 12-weeks aerobic exercise intervention
  Interventions: Behavioral: Aerobic exercise
- Control (No Intervention): Usual care, with recommendations for a healthy lifestyle.

INTERVENTIONS:
Behavioral: Aerobic exercise — 12-weeks aerobic exercise intervention based on the physical activity guidelines from the American College of Sports Medicine (≥150 min/week of moderate to vigorous [40-85% of the individual's heart rate reserve] exercise). Participants will perform the exercise on treadmills at the hospital. The volume and intensity of the exercise will progressively increase throughout the 12 weeks.
  Arms: Exercise

SUMMARY:
Patients with Systemic Lupus Erythematosus (SLE) have increased arterial stiffness, which leads to cardiovascular diseases (CVD) of arteriosclerotic origin, which are the main cause of mortality in these patients. Exercise is a modifiable factor that reduces cardiovascular mortality and associated risk factors in the general population. Preliminary studies suggest that exercise may improve endothelial function and lipid profile in patients with SLE. However, whether meeting the international physical activity guidelines from the American College of Sports Medicine (ACSM; i.e. ≥150 min / week of moderate to vigorous intensity physical activity) can improve arterial stiffness (subclinical atherosclerosis marker) and inflammation is unknown.

The primary aim of this study is to assess the effect of an exercise program based on meeting the ACSM physical activity guidelines on arterial stiffness and inflammation in patients with SLE.

The secondary aim is to assess the effect of an exercise program based on meeting the ACSM physical activity guidelines on endothelial function, oxidative stress, as well as other cardiometabolic risk factors, physical fitness, health-related quality of life, and other psychosocial outcomes.

Our hypothesis is that meeting the ACSM guidelines will improve arterial stiffness and inflammation in patients with SLE.

The study is a non-randomized clinical trial. To minimize selection bias, participants in the intervention and control groups will be matched by age, BMI, and disease activity (SLEDAI), which are important contributors to arterial stiffness.

DETAILED DESCRIPTION:
2. Design and Protocol Registration This non-randomized controlled trial was registered at clinicaltrials.gov [NCT03107442] on 11 April 2017, before the enrolment of participants started (i.e., on 12 April), and no deviations occurred regarding the primary outcome and the secondary outcomes analyzed here.

3. Setting and Eligibility Criteria Participants were recruited from the Systemic Autoimmune Diseases Unit of the "Virgen de las Nieves" and the "San Cecilio" University Hospitals. Women with a diagnosis of SLE according to the ACR criteria [26], a follow-up of 12 months, clinical and treatment stability during the previous six months, and not performing regular exercise (defined as 60 min/week of structured exercise) were included. Exclusion criteria were to have been under biological treatment in the previous six months or to need a prednisone dose of >10 mg/day; a background of CVD in the previous year; to present contraindications to perform exercise; other associated rheumatic conditions; pregnancy; active acute or chronic infection; neoplasms; acute renal failure; cardiac or pulmonary involvement; body mass index (BMI) >35; or not being able to read, understand, and sign written informed consent.

All participants received detailed information about the study procedures, and signed written informed consent. The Research Ethics Committee of Granada approved the protocol on 11 November 2016 (reference No.: 10/2016).

4. Procedures A telephone screening was conducted. Potentially eligible participants were invited to a personal screening and, if included, day 1 of the baseline examination was performed. The baseline examination comprised two assessment days. On day 1, pulse wave velocity (PWV) was assessed. Thereafter, cardiorespiratory fitness testing was performed, and socio-demographic and clinical information was collected. On day 2 (i.e., between two and four days after day 1), 8-h fasting blood samples were collected between 8:00 a.m. and 10:00 a.m. This article follows the TREND statement for improving the reporting of non-randomized experiments of behavioral and public health interventions (downloadable at EQUATOR Network: https://goo.gl/ZSyLrj; Supplementary Table S1) [27]. The funding source had no role in the study.

5. Methods 5.1. Interventions 5.1. 1. Exercise Group To maximize transparency and replicability, the exercise program described in this manuscript follows the Consensus on Exercise Reporting Template (CERT; Supplementary Table S2) [28]. The patients assigned to exercise performed two 75-min sessions per week during a total of 12 weeks (i.e., 24 sessions) of moderate to vigorous intensity aerobic exercise on a treadmill (BH, Serie i.RC12 Dual, Vitoria-Gasteiz, Spain) from 24 April to 14 July 2017. The sessions took place in a quiet room of the "Virgen de las Nieves" Hospital, Granada (Spain).

All sessions were performed in groups of a maximum of five persons (depending on the patients' schedule preferences) and were supervised by both exercise professionals with a degree in Sports Sciences and residents from the Internal Medicine Department.

Attendance at the sessions was registered daily and patients were contacted upon any missing session to ask for the reason and motivate them to replace it on an alternative day of the same week. Adherence to exercise is reported as the median attendance frequency and the proportion of patients attending >75% (i.e., 18 sessions; the minimum pre-defined attendance to assess efficacy) and >90% of the sessions. All the sessions began with a warm-up comprising 3-4 min of activation on the treadmill at about 35-40% of the heart rate reserve (HRR) and 3-4 min of active stretching of major muscle groups, and ended with a cool down phase of static stretching of major muscle groups and relaxation. Exercise was individually prescribed to represent moderate-to-vigorous intensity, with training intensity ranging from 40% to 75% of each patient's HRR. The maximum heart rate (HRmax) was estimated with the formula by Tanaka et al. (HRmax = 208 x (0.7 x age)) [29]. The training (or target) heart rate (tHR) was calculated with the formula tHR = HRrest + (%HRR). Heart rate was continuously monitored during all sessions (Polar V800, Kempele, Finland). We used the session rating of perceived exertion (RPE) as a measure of subjective training load [30], and the feeling scale to assess positive affective responses experienced before and after each session [31].

The starting level was specific for each individual according to her previous exercise experience and physical fitness. During the first half of the program, only continuous exercise was performed so that the patients got used to the treadmill and felt confident at increasing intensities. Continuous sessions comprised several bouts of exertion at constant intensity, followed by a couple of minutes of recovery (i.e., rest) to drink water. During month 2, there were alternated continuous and interval sessions, and at month 3, the patients undertook interval training sessions, where there were periods of lower and periods of higher intensity efforts followed by some minutes of rest for hydration (Table 1). The progression in volume and/or intensity was patient-limited and was undertaken by increasing the treadmill speed (first) or inclination according to the symptoms and perceived exertion. There were no home-based or non-exercise components within this intervention. However, if a participant was eventually not able to attend a particular session, we provided her with a heart rate monitor and allowed recovery of that session out of the Hospital (a total of seven sessions were recovered in this fashion). Finally, the exercise intensity progressions had to be slightly modified from the initial plan. For instance, several patients perceived a 5% HRR intensity increase (i.e., from one week to another) as very heavy and difficult-to-follow. Consequently, there were weeks in which exercise intensity increased by 2.5% instead of 5% (Table 1).

5.1.2. Control Group After the baseline evaluation, the SLE patients assigned to the (usual care) control group received verbal information about a healthy lifestyle, including physical activity guidelines and basic nutritional information.

5.2. Outcome Measures Primary Outcome Measure: Arterial Stiffness Arterial stiffness was assessed in a sitting position by PWV [9], using the Mobil-O-Graph® 24 h pulse wave analysis monitor (IEM GmbH, Stolberg, Germany), whose operation is based on oscillometry recorded by a blood pressure cuff placed on the brachial artery. The coefficient of variation (CV) of Mobil-O-Graph for consecutive PWV analyses is 3.4% and its intraclass correlation coefficient is 0.98 [0.96-0.99] [32]. This device has been largely shown to be valid and reliable for measuring PWV and central blood pressure in different populations [33,34], meets the accuracy requirements of the British Hypertension Society (BHS) standard [35], and can be recommended for clinical use [36].

Secondary Outcome Measures Blood Samples and Biochemical Analyses Fasting blood specimens for biochemical and immunological tests were collected and routinely processed by the central laboratory of our hospital. Among other measurements, they included lipids, insulin (BioRad, Marne-la-Coquette, France), and a routine biochemical profile. The homeostatic model assessment for insulin resistance (HOMA-IR) was calculated (HOMA-IR = glucose (mmol/L) insulin ( U/L)/22.5).

Inflammatory Markers Serum high-sensitivity CRP was assessed by an immunoturbidimetric method using the ARCHITECT cSystems (MULTIGENT CRP Vario assay); the limit of quantitation was 0.2 mg/L and the upper limit for normal serum was 5 mg/L (coefficient of variation <6%). Interleukin 6 and TNF-

, as well as myeloperoxidase (MPO; as marker of oxidative stress), were measured in plasma. Serum was initially separated by centrifugation and stored at 70 C.

Bioserum concentrations of IL-6/TNF- (pg/mL) and MPO (ng/mL) were measured by an immunoradiometric assay using commercial kits (MILLIPLEX MAP Kit Human High Sensitivity T Cell Magnetic Bead Panel (HSTMAG-28SK) and Human Cardiovascular Disease Magnetic Bead Panel 2 (HCVD2MAG-67K)), Millipore) following the manufacturer's instructions. Quantitative data were obtained by using the Luminex-200 system (Luminex Corporation, Austin, TX, USA), and data analysis was performed on XPonent 3.1 software (Austin, TX, USA). The detections limits were 0.73 pg/mL for IL-6, 0.43 pg/mL for TNF-a, and 0.024 ng/mL for MPO.

Cardiorespiratory Fitness Cardiorespiratory fitness was assessed with the Bruce submaximal treadmill protocol [37]. The test comprised five increasing workload stages of 3 min each (stage 1: 2.7 km/h and 10% inclination; stage 2: 4 km/h and 12% inclination; stage 3: 5.5 km/h and 14% inclination; stage 4: 6.8 km/h and 16% inclination; stage 5: 8 km/h and 18% inclination). The test concluded when the participant achieved 85% of the individual's HRmax, as estimated with the formula by Tanaka et al. [29]. As validated SLE-specific formulas to estimate VO2max are not available, we used the total time to reach 85% HRmax as the outcome of interest.

Other Measurements All participants filled out a socio-demographic and clinical data questionnaire. Height (cm) was measured using a height gauge, weight (kg) with a bioimpedance device (InBody R20, Biospace, Seoul, Korea), and body mass index (BMI) was calculated (kg/m2). Blood pressure was measured with Mobil-O-Graph (IEM GmbH, Stolberg, Germany) [36]. Disease activity was assessed through the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI, range 0-105 where a higher score indicates higher degree of disease activity). Physical activity was self-reported at baseline and at week 12 with the International Physical Activity Questionnaire [38].

Sample Size The sample size was calculated for the primary outcome (i.e., PWV). Ashor et al. found an average effect of aerobic exercise on PWV of 0.63 m/s in adults aged 18 years [21]. A total of 52 patients (26 per group) were needed to detect an effect of 0.63 (SD 0.75) m/s, with a power of 85% and an error of 0.05. Anticipating a maximum loss to follow-up of 15%, we aimed at recruiting a total of 60 patients.

Treatment Allocation and Blinding Randomization was not feasible because more than half of the patients who regularly attend the Autoimmune Disease Units lived far from the Hospital and were not able to attend twice per week in case of being randomized to exercise. Therefore, participants from the city of Granada were included in the exercise group and participants living outside Granada were included in the control group.

To minimize potential selection bias, we aimed to match the groups by age ( 2 years), BMI ( 1 kg/m2), and SLEDAI ( 1 unit). The data analyzer was blinded to the patient allocation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus (SLE) according to the American College of Rheumatology criteria (presenting at least 4 classification criteria).
* Follow-up of at least 12 months at our Unit.
* Clinical and treatment stability during the 6 months prior to the study.
* Not performing regular exercise (defined as < 60min/week of structured exercise)

Exclusion Criteria:

* Biological treatment in the previous 6 months or to need prednisone dosis >10 mg/day.
* Background of clinical cardiovascular disease in the last year.
* To present contraindications to perform exercise.
* Other associated rheumatic conditions.
* Pregnancy.
* Acute renal failure.
* Cardiac or pulmonary involvement.
* Body Mass Index > 35
* Not being able to read, understand and sign written informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José A. Vargas-Hitos, MD, Ph.D., Principal Investigator — Virgen de las Nieves University Hospital, Granada, Spain
Locations (1):
- Virgen de las Nieves University Hospital, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | Control
Started | 26 | 32
Completed | 18 | 28
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Control | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (15.1) | 44.8 (13.1) | 44.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 32 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 26 | 32 | 58
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (3.4) | 24.7 (5.6) | 25.2 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Stiffness
Description: Pulse wave velocity assessed with Mobil-OGraph ® 24h pulse wave analysis monitor (IEM GmbH, Stolberg, Germany)
Time Frame: value at 12 weeks minus value at baseline
Measure: Median (Standard Error); unit: m/s
Arm/Group | Exercise | Control
Number analyzed (Participants) | 22 | 28
m/s | -0.26 (0.14) | -0.22 (0.13)

2. Secondary Outcome: Markers of Inflammation
Description: High sensitivity C-Reactive Protein (hs-CRP)
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: mg/L
Arm/Group | Exercise | Control
Number analyzed (Participants) | 22 | 28
mg/L | 0.17 (0.59) | -0.24 (0.55)

3. Secondary Outcome: Glucose
Description: Blood glucose levels
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
mg/dL | -3.12 (0.69) | 4.47 (3.77)

4. Secondary Outcome: Insulin
Description: Blood insulin levels
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: microUI/mL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
microUI/mL | -0.32 (0.09) | 0.30 (0.16)

5. Secondary Outcome: Homeostasis Model Assessment of Insulin Resistance
Description: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: HOMA Index
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
HOMA Index | -0.1 (0.03) | 0.22 (0.07)

6. Secondary Outcome: Glycated Hemoglobin
Description: Glycated hemoglobin (HbA1c %) obtained from blood sample
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: percentage hemoglobin
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
percentage hemoglobin | -0.02 (0.003) | 0.10 (0.02)

7. Secondary Outcome: Lipid
Description: Triglycerides
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
mg/dL | -2.72 (1.86) | 3.5 (0.62)

8. Secondary Outcome: Cardiorespiratory Fitness
Description: Assessed by the modified Bruce Test on a treadmill. The test comprised five increasing workload stages of 3 min each (stage 1: 2.7 km/h and 10% inclination; stage 2: 4 km/h and 12% inclination; stage 3: 5.5 km/h and 14% inclination; stage 4: 6.8 km/h and 16% inclination; stage 5: 8 km/h and 18% inclination). The test concluded when the participant achieved 85% of the individual's HRmax
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
minutes | 2.622 (0.41) | 0.43 (0.45)

9. Secondary Outcome: Muscle Strength
Description: Assessed by isometric handgrip dynamometry (hand grip strength test [TKK 5401, Takei Scientific Instruments, Tokyo, Japan]
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
Kg | 0.91 (0.33) | 0.27 (0.07)

10. Secondary Outcome: Flexibility
Description: Assessed by the back scratch test (from the Senior Fitness Test battery)
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: cm
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
cm | -0.03 (0.13) | -2.66 (0.05)

11. Secondary Outcome: Waist and Hip Circumference
Description: Waist and hip circumferences (cm) and ratio
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: Waist to hip ratio
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
Waist to hip ratio | 0.03 (0.2) | 0.02 (0.006)

12. Secondary Outcome: BMI
Description: Body Mass Index
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
kg/m^2 | 0.3 (0.03) | 0.51 (0.10)

13. Secondary Outcome: Coagulation
Description: Fibrinogen in Blood
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
mg/dL | 29.23 (13.99) | 38.1 (10.03)

14. Secondary Outcome: Renal Function
Description: Creatinine in blood sample
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
mg/dL | 0.01 (0.10) | -0.08 (0.03)

15. Secondary Outcome: Health-related Quality of Life
Description: The Spanish version of the 36-item Short-Form Health Survey (SF-36) was used to assess HRQoL. This questionnaire is validated for patients with SLE and it assesses eight health dimensions that define two global domains: the physical and mental component scales (PCS and MCS, respectively). Only the global domains were used for the present work, which scores range from 0 (worst possible health status) to 100 (the best possible health status).
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: points
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
points | 3.82 (2.07) | 0.21 (1.63)

16. Secondary Outcome: Depression
Description: Assessed by the Beck Depression Inventory second edition (BDI-II). Depressive symptomatology was assessed through the Beck Depression Inventory-second edition (BDI-II) [41]. This questionnaire has been used extensively in research, including SLE . It is a 21-item self-report measure where, according to how patients felt during the past 2 weeks, each depressive symptom is rated from 0 (not present) to 3 (severe). The BDI-II provides an overall score (0-63) where higher score indicates higher depressive symptomatology.
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: score on a scale
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
score on a scale | -3.32 (1.74) | -1.32 (1.56)

17. Secondary Outcome: Fatigue
Description: Fatigue was assessed with the Multidimensional Fatigue Inventory (MFI), which is a well-established instrument previously used in SLE. This questionnaire includes 5 subscales of fatigue severity: general, physical, and mental fatigue as well as reduced activity, and reduced motivation. Each subscale consists of four items ranging from 4 to 20, with higher scores indicating greater fatigue on that subscale.
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
units on a scale | -3 (0.74) | -0.01 (0.66)

18. Secondary Outcome: Sleep Quality
Description: Sleep quality over the last month interval was assessed with the Pittsburg Sleep Quality Index (PSQI), a widely-used instrument in SLE. This questionnaire is composed of 19 questions addressing a variety of factors related to sleep quality. The sleep quality global score is the sum of all components, that ranges from 0 to 21, with higher scores indicating worse sleep quality.
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
units on a scale | -0.96 (0.84) | -0.32 (0.65)

19. Secondary Outcome: Sedentary Behavior
Description: Assessed by the Sedentary Behavior Questionnaire (SBQ). Assesses the amount of time spent on nine different behaviours.
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: min/week
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
min/week | 129 (3.67) | 105 (10.83)

20. Secondary Outcome: Adherence to the Mediterranean Diet
Description: Adherence to the Mediterranean diet was estimated using the Mediterranean Diet Score. It consists of 11 items including whole grains, fruits, vegetables, potatoes, legumes, fish, poultry, dairy products (such as cheese, yogurt, and milk), red meats and their derivatives, olive oil, and red wine. Based on the portions the patients had consumed, the foods were scored from 0 to 5 (according to their position in the Mediterranean Diet pyramid). Total score ranges from 0 to 55, where higher scores indicate higher adherence to the Mediterranean diet and greater diet quality.
Time Frame: Change from baseline to week 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
score on a scale | -1.61 (0.01) | 0.71 (0.04)

21. Secondary Outcome: Perceived Stress
Description: Assessed by the Perceived Stress Scale (PSS). Psychological stress was measured with the Perceived Stress Scale (PSS), a 14-item self-report global measure designed to assess the degree to which situations in one's life are appraised as stressful [35]. The PSS have shown to be a valid and reliable measure in patients with SLE [36]. According to how patients felt during the last month, each item is rated from 0 (never) to 4 (very often). The PSS provides a single overall score (0-56) where higher score represents greater perceived stress.
Time Frame: Change from baseline to week 12
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Exercise | Control
Number analyzed (Participants) | 26 | 32
units on a scale | -1.6 (1.13) | -1.2 (1.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 3 months.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/32
Other Adverse Events (participants affected / at risk) | 0/26 | 0/32

LIMITATIONS AND CAVEATS:
This study has several limitations. First, the final sample size was relatively small and was calculated to assess the between-group change in arterial stiffness as the primary trial outcome. Consequently, the power to detect significant between-group differences in the outcomes reported was checked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03107442/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03107442/ICF_001.pdf